CLINICAL TRIAL: NCT05189353
Title: The Importance of Ghrelin for Glucose Metabolism After Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Marie-Louise Dichman, MD, Ph.d.-student, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: H-21037442
Record Dates: First submitted 2021-12-28; First posted 2022-01-12 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Bariatric Surgery Candidate; Glucose Metabolism Disorders
Keywords: Ghrelin; Gastric sleeve; Glucose metabolism
MeSH Terms: conditions — Glucose Metabolism Disorders | interventions — Ghrelin

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastric sleeve operated (Experimental): 12 subjects with normal glucose tolerance (NGT) operated with SG minimum 12 month earlier
  Interventions: Other: Ghrelin; Other: Placebo
- Matched control group (Placebo Comparator): 12 weight-matched unoperated subjects with NGT
  Interventions: Other: Ghrelin; Other: Placebo

INTERVENTIONS:
Other: Ghrelin — Ghrelin infusion
Other: Placebo — Saline infusion

SUMMARY:
The overall aim is to delineate the contribution of ghrelin to glucose tolerance after sleeve gastrectomy. The hypothesis is that decreased concentration of ghrelin after SG is of importance for improved insulin secretion and glucose tolerance seen after SG. The expectation is therefore that infusion of ghrelin will impair insulin secretion and glucose tolerance compared with a control day without ghrelin infusion.

DETAILED DESCRIPTION:
Roux-en-Y gastric bypass (RYGB) and sleeve gastrectomy (SG) are bariatric procedures. Overwhelming evidence support bariatric surgery as the most effective treatment for severe obesity and related metabolic comorbidities, particularly type 2 diabetes mellitus.

The mechanisms of improved glycaemic control after SG are not fully understood and differ from those of RYGB. Interestingly, there is demonstrated a markedly lower secretion of the orexigenic hormone ghrelin after SG compared with both RYGB and unoperated obese controls. Hence, the decreased level of ghrelin could be of major importance in relation to the improved glucose tolerance after SG.

Ghrelin is secreted from the gastric mucosa in the fasting state and decreases in response to food intake. Administration of exogenous ghrelin reduces insulin sensitivity and glucose tolerance in healthy humans and contributes to hyperglycaemia. In accordance, ghrelin receptor knockout in mice improves glucose sensitivity and enhances glucose-stimulated insulin secretion.

On this background the investigators hypothesize that the markedly reduced secretion of ghrelin after SG could therefore be of particularly importance for the improved glucose tolerance after this procedure.

This present study is complementary to an on-going study in SG operated subjects, where the role of ghrelin for appetite and insulin secretion during a mixed meal followed by an ad libitum meal are investigated. In the present study the effect of ghrelin on insulin secretion and insulin sensitivity is thoroughly investigated using methods eliminating the effect of other hormones on glucose metabolism.

Ghrelin will be infused in physiological doses aiming for plasma concentration after SG resembling the pre-operative plasma concentrations.

Specific aim is to evaluate the effect of ghrelin on both alpha and beta cell function as well as on liver and peripheral insulin sensitivity in individuals with SG using matched controls. The subjects will be investigated with both glucose and glycerol tracers, IVGTT and a hyperinsulinemic euglycaemic clamp.

ELIGIBILITY:
Inclusion Criteria:

* Sleeve gastrectomy-operated > 12 months prior to inclusion
* Weight stable (+/- 3 kg during the last 3 months)
* Fasting glucose < 7,0 mmol/l / HbA1c < 48 mmol/mol pre- and postoperative
* Signed written informed consent

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Haemoglobin < 6,5 mM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
The difference in disposition index between the two study days with and without ghrelin in fusion in the SG operated group | 0-180 minutes
  The first phase insulin response will be related to the ambient insulin sensitivity by calculating the disposition index (FPIR x M-value).

SECONDARY OUTCOMES:
The difference in first phase insulin response (FPIR) between the two study days with and without ghrelin in fusion in the SG operated group | 0-10 minutes (IVGTT)
  Estimation of beta-cell function, calculated from insulin secretion rate using c-peptid and deconvolution from 0-10 min.
The difference in Insulin sensitivity (M-value) between the two study days with and without ghrelin in fusion in the SG operated group | 160-180 minutes (the end of the clamp)
  When a steady state is reached at the end of the clamp, the glucose infusion rate represents insulin-mediated glucose uptake by the body.

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Universitets Hospital, Hvidovre, Denmark